CLINICAL TRIAL: NCT00358449
Title: A Randomized, Double-blind, Parallel Group Clinical Trial to Assess Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenous Mepolizumab (SB240563)(0.55mg/kg, 2.5mg/kg or 10mg/kg) in Pediatric Subjects With Eosinophilic Esophagitis, Aged 2 to 17 Years (Study MEE103219)
Brief Title: Intravenous Mepolizumab In Children With Eosinophilic Esophagitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEE103219
Record Dates: First submitted 2006-07-27; First posted 2006-07-31 (Estimated); Results first posted 2016-03-10 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-06

CONDITIONS: Oesophagitis, Eosinophilic
Keywords: eosinophilic; mepolizumab; esophagitis
MeSH Terms: conditions — Esophagitis | interventions — mepolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Mepolizumab 0.55 mg/kg (Experimental): Participants received mepolizumab 0.55 milligrams (mg)/kilogram (kg) by intravenous (IV) infusion for 30 minutes on Day 1, Week 4 and Week 8.
  Interventions: Drug: mepolizumab
- Mepolizumab 2.5 mg/kg (Experimental): Participants received mepolizumab 2.5 mg/kg by IV infusion for 30 minutes on Day 1, Week 4 and Week 8.
  Interventions: Drug: mepolizumab
- Mepolizumab 10 mg/kg (Experimental): Participants received mepolizumab 10 mg/kg by IV infusion for 30 minutes on Day 1, Week 4 and Week 8.
  Interventions: Drug: mepolizumab

INTERVENTIONS:
Drug: mepolizumab — Participants received mepolizumab 0.55 milligrams (mg)/kilogram (kg), 2.5 mg/kg , or 10 mg/kg by intravenous (IV) infusion for 30 minutes on Day 1, Week 4 and Week 8.

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of intravenous mepolizumab in pediatric subjects with eosinophilic esophagitis.

ELIGIBILITY:
Inclusion Criteria:

* A subject will be eligible for inclusion in this study only if all of the following criteria apply. Inclusion criteria pertain to all subjects in both cohorts (treatment and observational) unless otherwise stated.
* The subject signs and dates a written assent form (age appropriate) and the parent/guardian signs and dates a written informed consent form prior to the initiation of any study-related activities, including discontinuation of any prohibited medications.
* Male or female subjects aged 2 to 17 years (from 2nd birthday up to and not including 18th birthday), who weigh <=84.9kg (males)/ <= 72.5 (females) and who have a BMI between 5 and 85% for age, who speak, read and write English as age appropriate and/or parent/guardian.

NOTE: If subject is within weight requirements but close to the upper or lower limits at screening and the investigator anticipates that during the study the subject's weight will change a become outside the weight requirements, the subject should be excluded from the study.

* To be eligible for entry in the treatment group of the study, a female subject is eligible to enter the study if she is: not pregnant or nursing; of non-childbearing potential. Non-childbearing potential is defined as a pre-menarcheal female who has not yet entered puberty as evidenced by lack of breast development (palpable glandular breast tissue); or a female who has documentation (medical report verification) of hysterectomy and/or bilateral oophorectomy; of childbearing potential. These females subjects must have a negative urine pregnancy test at the screening visit, and agree to consistent and correct use of one of the acceptable methods of birth control from at least the commencement of their last normal period prior to the first dose of study medication and to continue until the first normal period after treatment or after the Week 24 Follow-up visit, whichever is longest.
* The subject has a diagnosis of eosinophilic esophagitis and current evidence on biopsy of isolated eosinophilic esophagitis defined as:
* Peak esophageal eosinophil counts (highest count of eosinophils per HPF in at least one of all esophageal sites biopsied) of 20 or more eosinophils in a minimum of one HPF at 400X magnification on histology of esophageal biopsies from distal and mid-esophagus within two weeks of commencing study medication, as determined by the central histopathologist.
* Inadequate response to or intolerant of therapy for eosinophilic esophagitis
* The individual investigators will apply their clinical judgment to define whether a clinical response to therapy for eosinophilic esophagitis is inadequate. As guidance, inadequate response might consist of persistence under current or recent prior therapy, of symptoms of eosinophilic esophagitis such as eosinophilic esophagitis-related pain in stomach, chest or throat; regurgitation; vomiting; pain or difficulties associated with drinking fluids or nutritional supplements; or pain or difficulties associated with eating. An inadequate response might also consist of persistent eosinophilic infiltration of the esophagus, in the presence or in the absence of eosinophilic esophagitis-related symptoms.
* Similarly, the individual investigators will apply their clinical judgment to define whether a patient is intolerant to therapy. For guidance, intolerance to therapy for eosinophilic esophagitis may consist of undesirable side-effects of long-term therapy; or side-effects of long-term therapy that are difficult to manage; or marked non-compliance to therapy or rejection of therapy by the individual patient, or by the parent/guardian, which in the opinion of the investigator interferes with the patient's optimal disease management.
* The criteria used by the investigator to define inadequate response to or intolerance of therapy for eosinophilic esophagitis will be collected in the CRF.

Exclusion Criteria:

* A subject will not be eligible for inclusion in this study if any of the following criteria apply. Exclusion criteria pertain to all subjects in both cohorts (treatment and observational) unless otherwise stated.
* Current evidence of eosinophilic gastrointestinal enteropathy (EGID), other than eosinophilic esophagitis.
* Evidence of gastroesophageal reflux disease, or other causes of esophagitis which in the investigator's opinion is the predominant cause of the subject's esophageal eosinophilia so that the investigator's opinion is allowed.
* Current presence, or history of (anytime in the past): hypereosinophilic syndromes, collagen vascular disease, vasculitis, allergic drug reaction as the cause of the peripheral eosinophilia, graft-versus host disease, chronic idiopathic inflammatory bowel disorders (ulcerative colitis, Crohn's disease, chronic granulomatous disease).
* Current evidence, or history of celiac disease.
* Current evidence of active H. pylori infection.
* Abnormal 12-lead ECG at Screening which is clinically significant in the opinion of the investigator. Note that this exclusion criterion does not apply for subjects who are considered for enrollment in the observational cohort.
* Use or administration of any of the prohibited medications from Screening and throughout completion of Week 34 follow-up. Note that this exclusion criterion does not apply for subjects who are considered for enrollment in the observational cohort.
* Failure to remain on a stable dose of one (or more) permitted medication(s) for at least 1 month prior to the Screening visit and throughout completion of Week 24 follow-up assessments. Note that this exclusion criterion does not apply for subjects who are considered for enrollment in the observational cohort.
* Failure to remain on stable elemental diet or dietary manipulations for at least 3 months prior to the Screening Visit and throughout completion of Week 34 follow-up assessments. Note that this exclusion criterion does not apply for subjects who are considered for enrollment in the observational cohort.
* Known history of allergic reaction to previous antibody therapy.
* Any previous treatment with anti-hIL-5, anti-IgE monoclonal antibody or other biological agents.
* Use of an investigational drug within 30 days of entering the study. Note that this exclusion criterion does not apply for subjects who are considered for enrollment in the observational cohort.
* Exhibits evidence of renal disease or serum creatinine > 1.5 times upper limit of normal range (ULN). Note that this exclusion criterion does not apply for subjects who are considered for enrollment in the observational cohort.
* Exhibits evidence of hepatic disease, impairment or abnormal liver function test i.e. AST, ALT >1.5 times ULN, bilirubin >1.5 times ULN. Note that this exclusion criterion does not apply for subjects who are considered for enrollment in the observational cohort.
* Known evidence of the following infections/infestations: HIV, Hepatitis B or C, Bacterial infection, Parasitic infestation.
* History or suspicion of current drug abuse and alcohol abuse within the last 6 months.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2006-09-11 (Actual); Primary Completion 2008-11-25 (Actual); Study Completion 2008-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (28):
- United States (19):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Springfield, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Southfield, Michigan
  - GSK Investigational Site, Troy, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Sioux Falls, South Dakota
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Milwaukee, Wisconsin
- GSK Investigational Site, Brisbane, Queensland, Australia
- Canada (4):
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Montreal, Quebec
- United Kingdom (4):
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London
  - GSK Investigational Site, Sheffield
  - GSK Investigational Site, Watford

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Assa'ad AH, Gupta SK, Collins MH, Thomson M, Heath AT, Smith DA, Perschy TL, Jurgensen CH, Ortega HG, Aceves SS. An antibody against IL-5 reduces numbers of esophageal intraepithelial eosinophils in children with eosinophilic esophagitis. Gastroenterology. 2011 Nov;141(5):1593-604. doi: 10.1053/j.gastro.2011.07.044. Epub 2011 Aug 9. PMID 21835135
- [Derived] Wong ECL, Gleave AL, Marshall JK, Narula N. Predictors of histologic response to mepolizumab in pediatric eosinophilic esophagitis. Eur J Gastroenterol Hepatol. 2023 Oct 1;35(10):1131-1136. doi: 10.1097/MEG.0000000000002623. Epub 2023 Jul 31. PMID 37577798
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: MEE103219 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: MEE103219 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: MEE103219 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: MEE103219 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: MEE103219 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: MEE103219 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: MEE103219 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (par.) who met the eligibility criteria were randomized in to Treatment Cohort (TC) that consisted of a 2-week Screening Phase, a 12-week Treatment Phase, a 12-week Follow-up Phase and a 10-week Long term Follow-up Phase. Eligible par. who chose not to enter TC could be enrolled in an Observational Cohort to be followed for 24 weeks.
Pre-assignment Details: A total of 77 subjects participated in this study. Of this total, 59 par. were randomized into the TC to receive blinded study medication. An additional 18 subjects elected not to participate in the TC and were enrolled in the Observational Cohort. A total of 113 par. were screened for eligibility, of which 36 were screen failures.
Period: Overall Study
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Started | 19 | 20 | 20
Completed | 15 | 19 | 18
Not Completed | 4 | 1 | 2
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Steriod Inhaler was Increased | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.4 (4.28) | 10.5 (5.15) | 10.4 (4.66) | 10.4 (4.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 3 | 12
  Male | 16 | 14 | 17 | 47
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 0 | 1 | 2 | 3
  Asian - Central/South Asian Heritage | 0 | 0 | 1 | 1
  White - White/Caucasian/European Heritage | 18 | 19 | 17 | 54
  Unknown | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Events (AE), Any Serious Adverse Event (SAE) and Drug-related AE During Treatment Phase (TP) and Follow-up Phase (FP)
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event is defined as any untoward medical occurrence that, at any dose that Results in death, life-threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; a congenital anomaly/birth defect. Drug-related AE's were considered to have a reasonable possibility of being related to treatment by the investigator. AE, SAE and drug-related AEs are summarized by TP and FP.
Time Frame: From first dose of study treatment (Day 1) up to Follow-up Phase (Week 24)
Population: Intention-to-Treat (ITT) Population: all participants who gave informed consent, were randomized and received at least one dose of medication.
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Participants
  Any AE, TP | 18 | 15 | 18
  Any AE, FP | 15 | 9 | 10
  Drug-Related AE, TP | 6 | 4 | 3
  Drug-Related AE, FP | 3 | 0 | 0
  Any SAE, TP | 0 | 1 | 2
  Any SAE, FP | 0 | 0 | 1

2. Primary Outcome: Number of Participants With Indicated Biochemistry Parameters Falling Outside of Reference Range (RR) in Any Vist Post-Basline During Study Period.
Description: Blood samples were collected at Day 1, Weeks 4, 8, 12, 16, 20 and 24 to estimate the following biochemistry parameters: alanine amino transferase (ALT), aspartate amino transferase (AST), albumin (Ab), total protein (ToP), creatinine (Cr), total bilirubin (TB), calcium (Ca), bicarbonate (Bi), chloride (Cl), glucose (Glu), potassium (Pot), and sodium (Sod). Laboratory abnormalities outside the reference range (high and low values) at any time post baseline were presented. Any time post Baseline = all visits (including scheduled and unscheduled). If participant had given both high and low value at least once then participant is counted under both high and low category for this visit.
Time Frame: From first dose of study treatment (Day 1) up to Follow-up Phase (Week 24)
Population: ITT Population. Only those participants available at specified time points are analyzed (represented as n=X,X,X in the category titles).
Measure: Number; unit: Participants
Groups:
- Mepolizumab 0.55 mg/kg: Participants received mepolizumab 0.55 mg/kg by IV infusion for 30 minutes on Day 1, Week 4 and Week 8.
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Participants
  ALT - RR High, n=19 ,20, 20 | 3 | 0 | 3
  ALT - RR Low, n=19, 20, 20 | 1 | 0 | 1
  AST - RR High, n=19, 20, 20 | 5 | 4 | 7
  AST - RR Low, n=19, 20, 20 | 0 | 2 | 0
  Ab - RR High, n=19, 20, 20 | 5 | 1 | 2
  Ab - RR Low, n=19, 20, 20 | 4 | 3 | 5
  ToP - RR High, n=19, 20, 20 | 0 | 2 | 1
  ToP - RR Low, n=19, 20, 20 | 6 | 4 | 6
  Cr - RR High, n=19, 20, 20 | 2 | 4 | 3
  Cr - RR Low, n=19, 20, 20 | 3 | 3 | 4
  TB - RR High, n=19, 20, 20 | 0 | 0 | 0
  TB - RR Low, n=19, 20, 20 | 3 | 3 | 4
  Ca - RR High, n=19, 20, 20 | 4 | 7 | 7
  Ca - RR Low, n=19, 20, 20 | 2 | 0 | 0
  Bi - RR High, n=19, 20, 20 | 6 | 2 | 2
  Bi - RR Low, n=19, 20, 20 | 0 | 1 | 0
  Cl - RR High, n=19, 20, 20 | 1 | 1 | 1
  Cl - RR Low, n=19, 20, 20 | 1 | 0 | 0
  Glu - RR High, n=19, 20, 20 | 8 | 8 | 7
  Glu - RR Low, n=19, 20, 20 | 9 | 7 | 8
  Pot - RR High, n=19, 19, 20 | 1 | 1 | 0
  Pot - RR Low, n=19, 19, 20 | 1 | 0 | 0
  Sod - RR High, n=19, 20, 20 | 0 | 0 | 0
  Sod - RR Low, n=19, 20, 20 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Indicated Hematology Parameters Falling Outside of Reference Range (RR) in Any Vist Post-Basline During the Study Period.
Description: Blood samples were collected pre-infusion at Day 1, Week 4 and Week 8; and 24h and 72h post-infusion at Day 1, Week 4 and Week 8 time points and at Weeks 2, 6, 10, 12, 16, 20, 24, and 34 to estimate the following hematology parameters: basophils (Bas), percentage of basophils (% Bas), lymphocytes (Lym), percentage of Lym (% Lym), monocytes (Mon), percentage of Mon (% Mon), platelet count (PC), total neutrophils (TN), percentage of TN (% TN), white blood cell count (WBC), hematocrit (He), hemoglobin (Hg), and red blood cell count (RBC). Laboratory abnormalities outside the reference range (high and low values) at any time post baseline were presented. Any time post Baseline = all visits (including scheduled and unscheduled). If participant had given both high and low value at least once then participant is counted under both high and low category for this visit.
Time Frame: From first dose of study treatment (Day 1) up to Long-term Follow-up Phase (Week 34)
Population: ITT Population. Only those participants available at specified time points are analyzed.
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Participants
  Bas - RR High | 1 | 2 | 0
  Bas - RR Low | 0 | 0 | 0
  % Bas - RR High | 0 | 3 | 3
  % Bas - RR Low | 0 | 0 | 0
  Lym - RR High | 0 | 1 | 0
  Lym - RR Low | 1 | 0 | 0
  % Lym -RR High | 12 | 10 | 12
  % Lym -RR Low | 2 | 1 | 4
  Mon -RR High | 6 | 7 | 4
  Mon - RR Low | 3 | 4 | 5
  % Mon -RR High | 14 | 12 | 15
  % Mon -RR Low | 1 | 3 | 4
  PC - RR High | 3 | 4 | 3
  PC - RR Low | 1 | 2 | 0
  TN - RR High | 2 | 4 | 6
  TN - RR Low | 5 | 5 | 3
  % TN - RR High | 1 | 1 | 4
  % TN -RR Low | 15 | 11 | 13
  WBC - RR High | 2 | 5 | 4
  WBC - RR Low | 7 | 4 | 7
  He - RR High | 0 | 1 | 1
  He - RR Low | 6 | 6 | 5
  Hg - RR High | 0 | 0 | 1
  Hg - RR Low | 4 | 4 | 1
  RBC - RR High | 0 | 0 | 1
  RBC - RR Low | 4 | 7 | 7

4. Primary Outcome: Number of Participants With the Indicated Change From Baseline in ECG Findings at Any Time Post-Baseline
Description: 12-lead ECG assessments were obtained at the following time points: screening, and Weeks 4, 8 and 12.. Overall ECG findings were summarized using the worst case findings without regard to visits ie. "any time post Baseline". Change from Baseline in ECG findings were categorized as clinically significant change from Baseline; no clinically significant change from Baseline and not applicable.
Time Frame: Screening, Weeks 4, 8 and 12
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Participants
  Clinically significant change from | 1 | 0 | 0
  No clinically significant change from | 18 | 20 | 20
  Not applicable | 0 | 0 | 0

5. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at the Indicated Time Points
Description: SBP and DBP measurements were obtained at the following time points: screening, pre-infusion, 10 minutes (m), 30m, 1 hour (h), 2h post-infusion on Day 1, Week 4, Week 8; and Weeks 12, 16, 20 and 24. Screening value was considered as the Baseline value. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Screening, Day 1, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Millimeters of mercury (mmHg)
  SBP, Day 1 pre-infusion, n= 19, 20, 20 | 1.2 (10.65) | 3.4 (16.10) | 7.4 (14.09)
  SBP, Day 1, 10m, n= 19, 20, 19 | -3.2 (10.82) | 0.8 (12.16) | 4.8 (15.27)
  SBP, Day 1, 30m, n= 19, 20, 20 | -1.7 (11.94) | 1.6 (12.75) | 5.4 (15.53)
  SBP, Day 1, 1h, n= 19, 20, 20 | 1.1 (13.68) | 2.0 (13.45) | 3.6 (14.55)
  SBP, Day 1, 2h, n= 19, 20, 20 | -0.6 (10.32) | 2.8 (10.08) | 2.7 (15.92)
  SBP, Week 4 pre-infusion, n= 19, 20, 19 | 4.2 (8.74) | 0.2 (11.04) | 5.7 (12.67)
  SBP, Week 4, 10m, n= 19, 20, 19 | -1.7 (11.32) | -0.8 (15.93) | 3.2 (13.62)
  SBP, Week 4, 30m, n= 19, 19, 19 | 1.2 (10.71) | -4.1 (15.26) | 2.5 (16.33)
  SBP, Week 4, 1h, n= 19, 19, 20 | -1.6 (9.91) | -4.8 (12.69) | 4.2 (16.44)
  SBP, Week 4, 2h, n= 19, 19, 20 | -0.7 (8.69) | 0.5 (12.99) | 2.9 (15.79)
  SBP, Week 8 pre-infusion, n= 19, 20, 19 | -0.2 (11.18) | 1.2 (13.74) | 10.4 (13.08)
  SBP, Week 8, 10m, n= 19, 20, 19 | -1.7 (10.58) | -1.0 (17.12) | 3.3 (14.31)
  SBP, Week 8, 30m, n= 19, 19, 18 | -2.7 (10.29) | 0.8 (15.90) | 2.2 (15.89)
  SBP, Week 8, 1h, n= 19, 19, 17 | 1.2 (13.30) | -0.6 (14.18) | 8.7 (15.73)
  SBP, Week 8, 2h, n= 19, 18, 18 | 0.4 (12.97) | 0.3 (13.11) | 4.6 (14.41)
  SBP, Week 12, n= 18, 20, 20 | 1.2 (12.27) | 2.1 (15.37) | 12.1 (15.12)
  SBP, Week 16, n= 15, 19, 20 | -1.5 (10.33) | 2.3 (11.98) | 9.7 (18.97)
  SBP, Week 20, n= 15, 18, 18 | 0.7 (8.80) | 2.8 (14.96) | 13.1 (14.55)
  SBP, Week 24, n= 17, 20, 19 | 2.1 (9.23) | 2.5 (12.33) | 6.9 (15.13)
  DBP, Day 1 pre-infusion, n= 19, 20, 20 | -0.1 (8.81) | 2.0 (11.23) | 1.4 (9.36)
  DBP, Day 1, 10m, n= 19, 20, 19 | -1.5 (9.03) | -1.2 (11.37) | 2.1 (11.98)
  DBP, Day 1, 30m, n= 19, 20, 20 | -0.2 (7.93) | -1.2 (10.89) | -0.7 (12.11)
  DBP, Day 1, 1h, n= 19, 20, 20 | -1.7 (8.41) | -1.1 (10.94) | -2.4 (13.43)
  DBP, Day 1, 2h, n= 19, 20, 20 | -0.1 (7.39) | 1.5 (14.34) | -0.4 (12.96)
  DBP, Week 4 pre-infusion, n= 19, 20, 19 | -0.2 (7.79) | 1.3 (9.97) | 1.2 (11.46)
  DBP, Week 4, 10m, n= 19, 20, 19 | -1.5 (8.82) | -1.6 (11.97) | -0.3 (12.71)
  DBP, Week 4, 30m, n= 19, 19, 19 | -0.4 (10.31) | -1.7 (11.51) | -0.9 (12.10)
  DBP, Week 4, 1h, n= 19, 19, 20 | -2.0 (7.54) | -3.9 (9.14) | 1.5 (13.45)
  DBP, Week 4, 2h, n= 19, 19, 20 | 0.8 (10.21) | 1.6 (9.42) | 0.5 (14.38)
  DBP, Week 8 pre-infusion, n= 19, 20, 19 | 0.9 (7.92) | -0.7 (9.50) | 4.1 (12.01)
  DBP, Week 8, 10m, n= 19, 20, 19 | -1.7 (7.72) | -2.2 (11.28) | 1.7 (15.01)
  DBP, Week 8, 30m, n= 19, 19, 18 | -2.2 (9.08) | -0.4 (13.68) | -3.3 (14.15)
  DBP, Week 8, 1h, n= 19, 19, 17 | -2.3 (11.44) | -1.1 (11.97) | 0.1 (14.61)
  DBP, Week 8, 2h, n= 19, 18, 18 | -4.4 (9.66) | -0.9 (11.69) | -1.2 (13.53)
  DBP, Week 12, n= 18, 20, 20 | -1.9 (9.09) | -1.8 (5.21) | 5.5 (14.48)
  DBP, Week 16, n= 15, 19, 20 | 0.6 (10.06) | 3.2 (12.39) | 3.1 (12.33)
  DBP, Week 20, n= 15, 18, 18 | -2.5 (7.90) | 3.4 (10.05) | 3.3 (11.26)
  DBP, Week 24, n= 17, 20, 19 | -0.2 (9.26) | 2.3 (10.02) | 3.5 (8.42)

6. Primary Outcome: Change From Baseline in Heart Rate at the Indicated Time Points
Description: Heart rate measurements were obtained at the following time points: Screening, pre-infusion, 10m, 30m, 1h, 2h post-infusion on Day 1, Week 4, Week 8; and Weeks 12, 16, 20 and 24. Screening value was considered as the Baseline value. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Screening, Day 1, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Beats per minutes
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Beats per minutes
  Day 1 pre-infusion, n= 19, 20, 20 | 0.7 (10.29) | 4.0 (12.21) | 2.3 (10.76)
  Day 1, 10m, n= 19, 20, 19 | -3.6 (9.39) | 1.7 (15.36) | 0.1 (12.34)
  Day 1, 30m, n= 19, 20, 20 | -2.5 (13.02) | 3.5 (14.36) | 1.9 (11.56)
  Day 1, 1h, n= 19, 20, 20 | -4.2 (11.51) | 3.0 (13.56) | 0.9 (15.40)
  Day 1, 2h, n= 19, 20, 20 | 1.6 (11.31) | 4.7 (15.08) | -0.5 (12.53)
  Week 4 pre-infusion, n= 19, 20, 19 | 0.4 (19.19) | 2.0 (13.13) | 1.4 (14.56)
  Week 4, 10m, n= 19, 20, 19 | -0.9 (13.56) | -1.6 (11.93) | -4.8 (14.83)
  Week 4, 30m, n= 19, 19, 19 | -1.4 (15.36) | -4.3 (13.67) | -4.0 (9.71)
  Week 4, 1h, n= 19, 19, 20 | -4.9 (14.08) | -1.8 (12.88) | -2.2 (15.10)
  Week 4, 2h, n= 19, 19, 20 | -3.3 (14.63) | -0.8 (10.58) | -5.3 (14.26)
  Week 8 pre-infusion, n= 19, 20, 19 | -3.1 (12.71) | 1.5 (12.15) | 7.1 (21.13)
  Week 8, 10m, n= 19, 20, 19 | -2.8 (11.69) | -4.6 (15.37) | 0.1 (16.18)
  Week 8, 30m, n= 19, 19, 18 | -3.8 (12.19) | -2.7 (9.52) | -2.1 (18.73)
  Week 8, 1h, n= 19, 19, 17 | -6.2 (10.73) | 0.3 (11.09) | 0.9 (12.46)
  Week 8, 2h, n= 19, 18, 18 | -5.4 (11.14) | 5.7 (10.33) | -0.3 (12.30)
  Week 12, n= 18, 20, 20 | -1.8 (13.58) | 0.3 (13.05) | 1.1 (14.37)
  Week 16, n= 15, 19, 20 | -7.1 (14.64) | 6.9 (13.12) | 2.9 (12.62)
  Week 20, n= 15, 18, 18 | -6.1 (17.40) | 7.8 (14.81) | 1.7 (15.50)
  Week 24, n= 17, 20, 19 | -2.1 (13.03) | 0.5 (13.43) | -0.4 (13.41)

7. Primary Outcome: Change From Baseline in Temperature at the Indicated Time Points
Description: Temperature measurements were obtained at the following time points: Screening, Day 1, and Weeks 4, 8, 12, 16, 20 and 24. Screening value was considered as the Baseline value. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Screening, Day 1, Weeks 4, 8, 12, 16, 20 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Degree Celsius (°C)
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Degree Celsius (°C)
  Day 1, n=19, 20, 20 | -0.18 (0.472) | 0.01 (0.824) | -0.07 (0.758)
  Week 4, n=19, 20, 20 | -0.44 (1.023) | -0.30 (0.614) | -0.14 (0.909)
  Week 8, n=19, 20, 19 | -0.44 (0.490) | -0.13 (0.696) | -0.06 (0.819)
  Week 12, n=18, 20, 20 | 0.03 (0.661) | -0.09 (0.671) | -0.08 (0.914)
  Week 16, n=15, 17, 20 | -0.01 (0.518) | 0.05 (0.491) | 0.02 (0.753)
  Week 20, n=15, 18, 18 | 0.00 (0.626) | -0.12 (0.696) | -0.12 (0.644)
  Week 24, n=17, 20, 19 | -0.11 (0.506) | -0.31 (0.668) | -0.12 (0.826)

8. Primary Outcome: Number of Participants With Positive and Negative Anti-mepolizumab Antibody Results at Any Visit and Repeat Visit.
Description: Blood samples for testing anti-mepolizumab antibodies were collected on Day 1, Week 4 and 8 Infusion Visit (before the IV infusion) and at Week 12, 24 and 34 Week follow-up visits. The presence of anti-human mepolizumab antibodies was assessed using an immunoelectrochemiluminescent (ECL) assay. To address transient positive results, an assessment of repeated results were made. For any visit category: results were considered as positive if it was positive at any visit during the study, and results were considered as negative if it were negative at all visits during the study. For repeat visit category: results were considered as postive if the result was positive at >1 visit, and results were considered as negative if the result was negative at all visits or was positive at only one visit.
Time Frame: Day 1, Weeks 4, 8, 12, 24, and 34
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Participants
  Any Visit- ECL Screening Positive | 15 | 15 | 16
  Any Visit- ECL Screening Negative | 4 | 5 | 4
  Repeat Visit-ECL Screening Positive | 13 | 5 | 7
  Repeat Visit-ECL Screening Negative | 6 | 15 | 13

9. Primary Outcome: Number of Participants Achieving a Reduction in Peak Esophageal Eosinophil Count to < 5 Cells Per High Power Field (HPF) at Week 12
Description: A responder was defined as a participant achieving a reduction in esophageal eosinophils to <5 cells per HPF as the highest count of eosinophils per HPF in all the esophageal sites biopsied at Week 12, confirmed by biopsy at Week 12 or at an early withdrawal visit prior to Week 12. A worst case (WC) approach was considered, if a particiapant withdrew prematurely : If a particiapnt dropped out of the study without having a biopsy taken, due to lack of efficacy or an adverse event, their response was imputed as not achieved. Participants who withdrew, without a biopsy, for other reasons (e.g. lost to follow-up) were considered non-evaluable for the primary analysis. For participants who withdrew early from the study and had a biopsy, the biopsy was used to determine their response.
Time Frame: Week 12
Population: ITT Population-WC
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 17 | 20 | 20
Participants | 3 | 2 | 0
Statistical Analysis 1: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.865, Regression, Logistic; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.04 to 5.44]
Statistical Analysis 2: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.190, Regression, Logistic; Odds Ratio (OR) = 0.21, 95% CI 2-sided [0.01 to 2.07]

10. Primary Outcome: Central (V1), Periperial (V2) and Steady-State (Vss) Volume of Distribution of Mepolizumab
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug is uniformly distributed to produce the desired plasma concentration of a drug. Central volume of distribution is a hypothetical volume into which a drug initially distributes upon administration. Peripheral volume of distribution is the sum of all tissue spaces outside the central compartment. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state. Blood samples were obtained at pre-infusion and 5m, 2h, 24h, 72-96h post-infusion at Day 1, Weeks 4, 8; and Weeks 2, 6 10, 12, 16, 20, 24 and 34 from each participant to estimate central (V1) and periperial (V2) and Steady State (Vss) volume of distribution of mepolizumab.
Time Frame: Day 1, Weeks 2, 4, 6, 8, 10, 12, 16, 20, 24, and 34
Population: Pharmacokinetic Population: all participants who received study medication and for whom mepolizumab sample was obtained and analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Liters
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Liters
  Central volume of distribution (V1) | 2.00 [1.62 to 2.48] | 2.29 [1.76 to 2.98] | 2.14 [1.60 to 2.88]
  Peripheral Volume of distribution (V2) | 1.36 [1.10 to 1.69] | 1.55 [1.19 to 2.03] | 1.46 [1.09 to 1.96]
  Steady-State Volume of distribution (Vss) | 3.37 [2.72 to 4.17] | 3.84 [2.95 to 5.00] | 3.60 [2.68 to 4.84]

11. Primary Outcome: Plasma Clearance (CL) of Mepolizumab
Description: Clearance is defined as the removal of drug from a volume of plasma in a given unit of time (drug loss from the body). Blood samples were obtained at pre-infusion and 5m, 2h, 24h, 72-96h post-infusion at Day 1, Weeks 4, 8; and Weeks 2, 6 10, 12, 16, 20, 24 and 34 from each participant to estimate plasma clearance of mepolizumab.
Time Frame: Day 1, Weeks 2, 4, 6, 8, 10, 12, 16, 20, 24, and 34
Population: Pharmacokinetic Population
Measure: Geometric Mean (95% Confidence Interval); unit: Liters per Day (L/day)
Groups:
- Mepolizumab 0.55/ 2.5/ 10 mg/kg: Participants received mepolizumab 0.55 mg/kg by IV infusion for 30 minutes on Day 1, Week 4 and Week 8.
Arm/Group | Mepolizumab 0.55/ 2.5/ 10 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Liters per Day (L/day) | 0.14 [0.11 to 0.18] | 0.15 [0.12 to 0.19] | 0.14 [0.12 to 0.18]

12. Secondary Outcome: Change From Baseline in Pain in Stomach Severity Scores
Description: Par.and/or parent/guardian recorded daily symptoms of eosinophilic esophagitis on a hand held personal digital assistant (electronic diary) during the Screening Phase, TP, and FP. A severity score of 0 was assigned for days on which pain in stomach was not experienced. If pain in stomach was reported, severity of pain was assessed as: 1=hurt a little, 2=hurt somewhat, 3=hurt quite a bit, and 4=hurt a whole lot. The average pain severity for the interval (Baseline, Weeks 9-12, Weeks 21-24) was calculated as the sum of the pain severity scores for that interval (including days assigned as 0) divided by the number of days in the interval. Screening phase was considered as the Baseline interval. Change from Baseline was calculated as the value for that interval minus the value for the Baseline interval. Analysis was performed using parametric Analysis of Covariance (ANCOVA) models with terms for the relevant Baseline score, treatment group, age group and treatment by age group interaction
Time Frame: Screening, Weeks 9-12 and Weeks 21-24
Population: ITT Population. The observed case (OC) datasets with incorrect questionnaires excluded were used for the analysis. Only those participants available at specified time points are analyzed (represented as n=X,X,X in the category titles).
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Scores on a scale
  Weeks 9-12, n= 15,18,13 | -0.277 [-0.617 to 0.062] | -0.149 [-0.412 to 0.115] | -0.157 [-0.458 to 0.144]
  Weeks 21-24, n=13,16,11 | -0.479 [-0.942 to 0.016] | -0.144 [-0.467 to 0.178] | -0.268 [-0.677 to 0.142]
Statistical Analysis 1: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.551, ANCOVA; Mean Difference (Final Values) = 0.128, 95% CI 2-sided [-0.303 to 0.560] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 2: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.593, ANCOVA; Mean Difference (Final Values) = 0.120, 95% CI [-0.331 to 0.572] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 3: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.239, ANCOVA; Mean Difference (Final Values) = 0.334, 95% CI 2-sided [-0.232 to 0.901] — P-value, 95% CI, and estimated value are presented for Weeks 21-24
Statistical Analysis 4: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.488, ANCOVA; Mean Difference (Final Values) = 0.211, 95% CI 2-sided [-0.401 to 0.823] — P-value, 95% CI, and estimated value are presented for Weeks 21-24

13. Secondary Outcome: Change From Baseline in Pain in Chest/Throat Severity Scores
Description: Par. and/or parent/guardian recorded daily symptoms of eosinophilic esophagitis on a hand held personal digital assistant (electronic diary) during the Screening Phase, TP, and FP. A severity score of 0 was assigned for days on which pain in chest/throat was not experienced. If pain in chest/throat was reported, severity of pain was assessed as: 1=hurt a little, 2=hurt somewhat, 3=hurt quite a bit, and 4=hurt a whole lot. The average pain severity for the interval (Baseline, Weeks 9-12, Weeks 21-24) was calculated as the sum of the pain severity scores for that interval (including days assigned as 0) divided by the number of days in the interval. Screening phase was considered as the Baseline interval. Change from Baseline was calculated as the value for that interval minus the value for the Baseline interval. Analysis was performed using parametric ANCOVA models with terms for the relevant Baseline score, treatment group, age group and treatment by age group interaction.
Time Frame: Screening, Weeks 9-12 and Weeks 21-24
Population: ITT Population. The OC datasets with incorrect questionnaires excluded were used for the analysis. Only those participants available at specified time points are analyzed (represented as n=X,X,X in the category titles).
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Scores on a scale
  Weeks 9-12, n=15,18,13 | -0.419 [-0.796 to -0.042] | -0.063 [-0.356 to 0.230] | -0.049 [-0.382 to 0.285]
  Weeks 21-24, n=13,16,11 | -0.524 [-0.943 to -0.105] | -0.091 [-0.385 to 0.202] | -0.181 [-0.551 to 0.188]
Statistical Analysis 1: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.139, ANCOVA; Mean Difference (Final Values) = 0.356, 95% CI 2-sided [-0.121 to 0.833] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 2: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.145, ANCOVA; Mean Difference (Final Values) = 0.371, 95% CI [-0.133 to 0.874] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 3: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.095, ANCOVA; Mean Difference (Final Values) = 0.433, 95% CI 2-sided [-0.080 to 0.946] — P-value, 95% CI, and estimated value are presented for Weeks 21-24
Statistical Analysis 4: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.219, ANCOVA; Mean Difference (Final Values) = 0.343, 95% CI 2-sided [-0.214 to 0.899] — P-value, 95% CI, and estimated value are presented for Weeks 21-24

14. Secondary Outcome: Change From Baseline in Percentage of Days With Pain in Stomach
Description: The percentage of days with the symptom of pain in stomach during each analysis interval (Baseline, Weeks 9-12 and Weeks 21-24) was calculated as the number of days the symptom was experienced divided by the number of days in the analysis interval, and presented as a percentage (ie, the proportion X 100%). Screening phase was considered as Baseline interval. Change from Baseline for each analysis interval was calculated as the value for that interval minus the value for the Baseline interval. Analysis was performed using parametric ANCOVA model with terms for Baseline score, treatment group, age group and treatment by age group interaction. The OC datasets with incorrect questionnaires excluded were used for the analysis.
Time Frame: Screening, Weeks 9-12 and Weeks 21-24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of days
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Percentage of days
  Weeks 9-12, n=15,18,13 | -14.02 [-25.93 to -2.12] | -12.44 [-21.66 to -3.21] | -10.11 [-20.70 to 0.48]
  Weeks 21-24, n=13,16,11 | -22.80 [-42.20 to -3.39] | -10.97 [-24.62 to 2.68] | -7.70 [-25.17 to 9.77]
Statistical Analysis 1: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.832, ANCOVA; Mean Difference (Final Values) = 1.59, 95% CI 2-sided [-13.47 to 16.65] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 2: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.622, ANCOVA; Mean Difference (Final Values) = 3.92, 95% CI 2-sided [-12.01 to 19.84] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 3: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.317, ANCOVA; Mean Difference (Final Values) = 11.83, 95% CI 2-sided [-11.86 to 35.52] — P-value, 95% CI, and estimated value are presented for Weeks 21-24
Statistical Analysis 4: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.246, ANCOVA; Mean Difference (Final Values) = 15.10, 95% CI 2-sided [-10.91 to 41.11] — P-value, 95% CI, and estimated value are presented for Weeks 21-24

15. Secondary Outcome: Change From Baseline in Percentage of Days With Pain in Chest/Throat
Description: The percentage of days with the symptom of pain in chest/throat during each analysis interval (Baseline, Weeks 9-12 and Weeks 21-24) was calculated as the number of days the symptom was experienced divided by the number of days in the analysis interval, and presented as a percentage (ie, the proportion X 100%). Screening phase was considered as Baseline interval. Change from Baseline for each analysis interval was calculated as the value for that interval minus the value for the Baseline interval. Analysis was performed using parametric ANCOVA model with terms for Baseline score, treatment group, age group and treatment by age group interaction. The OC datasets with incorrect questionnaires excluded were used for the analysis.
Time Frame: Screening, Weeks 9-12 and Weeks 21-24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of days
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Percentage of days
  Weeks 9-12, n=15,18,13 | -24.37 [-39.34 to -9.40] | -5.09 [-16.64 to 6.47] | -10.16 [-23.38 to 3.06]
  Weeks 21-24, n=13,16,11 | -27.12 [-43.32 to 10.93] | -9.43 [-20.80 to 1.94] | -6.01 [-20.34 to 8.32]
Statistical Analysis 1: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.046, ANCOVA; Mean Difference (Final Values) = 19.28, 95% CI 2-sided [0.39 to 38.18] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 2: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.160, ANCOVA; Mean Difference (Final Values) = 14.21, 95% CI 2-sided [-5.83 to 34.25] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 3: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.078, ANCOVA; Mean Difference (Final Values) = 17.69, 95% CI 2-sided [-2.10 to 37.48] — P-value, 95% CI, and estimated value are presented for Weeks 21-24
Statistical Analysis 4: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.055, ANCOVA; Mean Difference (Final Values) = 21.11, 95% CI 2-sided [-0.51 to 42.74] — P-value, 95% CI, and estimated value are presented for Weeks 21-24

16. Secondary Outcome: Change From Baseline in Regurgitation Bothersome Scores
Description: Par. and/or parent/guardian recorded daily symptoms of eosinophilic esophagitis on a hand held personal digital assistant (electronic diary) during the Screening Phase, TP, and FP. A score of 0 was assigned for days on which the symptom regurgitation was not experienced. The days regurgitation experienced, the amount the symptom bothered the Par. was assessed as 1=not bothered at all, 2=bothered a little, 3=somewhat bothered, 4=bothered quite a bit, 5=bothered a whole lot. The average pain severity for the interval (Baseline, Weeks 9-12, Weeks 21-24) was calculated as the sum of the pain severity scores for that interval (including days assigned as 0) divided by the number of days in the interval. Screening phase was considered as Baseline interval. Change from Baseline was calculated as the value for that interval minus the value for the Baseline interval. Analysis was performed using parametric ANCOVA models with terms for Baseline score, treatment group, age group interactions
Time Frame: Screening, Weeks 9-12 and Weeks 21-24
Population: ITT Population. The OC datasets with incorrect questionnaires excluded were the primary analysis. Only those participants available at specified time points are analyzed (represented as n=X,X,X in the category titles).
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Scores on a scale
  Weeks 9-12, n=15,18,13 | -0.307 [-0.741 to 0.128] | 0.017 [-0.320 to 0.354] | -0.047 [-0.431 to 0.337]
  Weeks 21-24, n=13,16,10 | -0.387 [-0.939 to 0.164] | -0.034 [-0.420 to 0.351] | -0.563 [-1.127 to 0.00]
Statistical Analysis 1: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.241, ANCOVA; Mean Difference (Final Values) = 0.324, 95% CI 2-sided [-0.226 to 0.873] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 2: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.371, ANCOVA; Mean Difference (Final Values) = 0.260, 95% CI 2-sided [-0.320 to 0.839] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 3: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.291, ANCOVA; Mean Difference (Final Values) = 0.353, 95% CI 2-sided [-0.317 to 1.023] — P-value, 95% CI, and estimated value are presented for Weeks 21-24
Statistical Analysis 4: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.653, ANCOVA; Mean Difference (Final Values) = -0.176, 95% CI 2-sided [-0.965 to 0.614] — P-value, 95% CI, and estimated value are presented for Weeks 21-24

17. Secondary Outcome: Change From Baseline in Percentage of Days With Regurgitation Bothersome Scores
Description: The percentage of days with the symptom of pain in regurgitation bothersome during each analysis interval (Baseline, Weeks 9-12 and Weeks 21-24) was calculated as the number of days the symptom was experienced divided by the number of days in the analysis interval, and presented as a percentage (ie, the proportion X 100%). Screening phase was considered as Baseline interval. Change from Baseline for each analysis interval was calculated as the value for that interval minus the value for the Baseline interval. Analysis was performed using parametric ANCOVA model with terms for Baseline score, treatment group, age group and treatment by age group interaction. The OC datasets with incorrect questionnaires excluded were used for the analysis.
Time Frame: Screening, Weeks 9-12 and Weeks 21-24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of days
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Percentage of days
  Weeks 9-12, n=15,18,13 | -10.26 [-24.44 to 3.91] | 3.80 [-7.32 to 14.93] | -4.64 [-17.15 to 7.88]
  Weeks 21-24, n=13,16,10 | -13.77 [-31.43 to 3.90] | 2.28 [-10.46 to 15.01] | -19.19 [-37.34 to -1.05]
Statistical Analysis 1: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.123, ANCOVA; Mean Difference (Final Values) = 14.06, 95% CI 2-sided [-4.00 to 32.13] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 2: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.551, ANCOVA; Mean Difference (Final Values) = 5.62, 95% CI 2-sided [-13.29 to 24.54] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 3: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.141, ANCOVA; Mean Difference (Final Values) = 16.04, 95% CI 2-sided [-5.61 to 37.70] — P-value, 95% CI, and estimated value are presented for Weeks 21-24
Statistical Analysis 4: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.666, ANCOVA; Mean Difference (Final Values) = -5.42, 95% CI 2-sided [-30.74 to 19.90] — P-value, 95% CI, and estimated value are presented for Weeks 21-24

18. Secondary Outcome: Change From Baseline in Frequency of Vomiting
Description: Par. and/or parent/guardian recorded daily symptoms of eosinophilic esophagitis on a hand held personal digital assistant (electronic diary) during the Screening Phase, TP, and FP. A participant vomiting any time was counted as one episode of vomiting, irrespective of how close they are to each other. The daily frequency of vomiting was calculated as the total number of times the participant vomited during the interval divided by the number of days in the interval. Screening phase was considered as Baseline interval. Change from Baseline was calculated as the value for that interval minus the value for the Baseline interval. Analysis was performed using parametric ANCOVA models with terms for the relevant Baseline score, treatment group, age group and treatment by age group interaction.
Time Frame: Screening, Weeks 9-12 and Weeks 21-24
Population: as for outcome 13
Measure: Least Squares Mean (95% Confidence Interval); unit: Occurrences of vomiting per day
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Occurrences of vomiting per day
  Weeks 9-12, n=15, 18, 13 | -0.048 [-0.296 to 0.199] | 0.040 [-0.149 to 0.229] | -0.060 [-0.281 to 0.161]
  Weeks 21-24, n=13, 16, 11 | -0.009 [-0.166 to 0.148] | -0.004 [-0.114 to 0.106] | 0.096 [-0.042 to 0.234]
Statistical Analysis 1: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.572, ANCOVA; Mean Difference (Final Values) = 0.088, 95% CI 2-sided [-0.224 to 0.400] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 2: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.942, ANCOVA; Mean Difference (Final Values) = -0.012, 95% CI 2-sided [-0.350 to 0.326] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 3: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.960, ANCOVA; Mean Difference (Final Values) = 0.005, 95% CI 2-sided [-0.188 to 0.197] — P-value, 95% CI, and estimated value are presented for Weeks 21-24
Statistical Analysis 4: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.317, ANCOVA; Mean Difference (Final Values) = 0.105, 95% CI 2-sided [-0.105 to 0.315] — P-value, 95% CI, and estimated value are presented for Weeks 21-24

19. Secondary Outcome: Change From Baseline in Percentage of Days With Vomiting
Description: The percentage of days with the symptom of vomiting during each analysis interval (Baseline, Weeks 9-12 and Weeks 21-24) was calculated as the number of days the symptom was experienced divided by the number of days in the analysis interval, and presented as a percentage (ie, the proportion X 100%). Screening phase was considered as Baseline interval. Change from Baseline for each analysis interval was calculated as the value for that interval minus the value for the Baseline interval. Analysis was performed using parametric ANCOVA model with terms for Baseline score, treatment group, age group and treatment by age group interaction. The OC datasets with incorrect questionnaires excluded were used for the analysis.
Time Frame: Screening, Weeks 9-12 and Weeks 21-24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of days
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Percentage of days
  Weeks 9-12, n=15,18,13 | -2.40 [-6.58 to 1.77] | -3.54 [-6.74 to -0.34] | -4.56 [-8.32 to -0.80]
  Weeks 21-24, n=13,16,11 | 1.62 [-4.43 to 7.67] | -2.98 [-7.22 to 1.27] | 1.11 [-4.24 to 6.45]
Statistical Analysis 1: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.666, ANCOVA; Mean Difference (Final Values) = -1.13, 95% CI 2-sided [-6.39 to 4.12] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 2: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.450, ANCOVA; Mean Difference (Final Values) = -2.16, 95% CI 2-sided [-7.87 to 3.56] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 3: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.215, ANCOVA; Mean Difference (Final Values) = -4.60, 95% CI 2-sided [-12.00 to 2.81] — P-value, 95% CI, and estimated value are presented for Weeks 21-24
Statistical Analysis 4: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.898, ANCOVA; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-8.61 to 7.58] — P-value, 95% CI, and estimated value are presented for Weeks 21-24

20. Secondary Outcome: Change From Baseline in Daily Degree of Difficulty With Drinking
Description: Par. and/or parent/guardian recorded daily symptoms of eosinophilic esophagitis on a hand held personal digital assistant (electronic diary) during the Screening Phase, TP, and FP. A score of 6 was assigned days the participant did not drink. The amount of difficulty with drinking was assessed as 1=no difficulty, 2=a little difficulty, 3=some difficulty, 4=quite a bit of difficulty, 5=a whole lot of difficulty. The average difficulty for the interval (Baseline, Weeks 9-12, Weeks 21-24) was calculated as the sum of the drinking difficulty scores for that interval (including days assigned as 6) divided by the number of days in the interval. Screening phase was considered as Baseline interval. Change from Baseline was calculated as the value for that interval minus the value for the baseline interval. Analysis was performed using parametric ANCOVA models with terms for the relevant Baseline score, treatment group, age group and treatment by age group interaction.
Time Frame: Screening, Weeks 9-12 and Weeks 21-24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Scores on a Scale
  Weeks 9-12, n=15,18,13 | 0.008 [-0.193 to 0.208] | 0.046 [-0.110 to 0.202] | -0.152 [-0.329 to 0.026]
  Weeks 21-24, n=13,16,11 | -0.137 [-0.420 to 0.145] | -0.049 [-0.245 to 0.147] | -0.070 [-0.315 to 0.175]
Statistical Analysis 1: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.762, ANCOVA; Mean Difference (Final Values) = 0.038, 95% CI 2-sided [-0.217 to 0.294] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 2: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.235, ANCOVA; Mean Difference (Final Values) = -0.159, 95% CI 2-sided [-0.426 to 0.108] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 3: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.607, ANCOVA; Mean Difference (Final Values) = 0.089, 95% CI 2-sided [-0.259 to 0.436] — P-value, 95% CI, and estimated value are presented for Weeks 21-24
Statistical Analysis 4: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.716, ANCOVA; Mean Difference (Final Values) = 0.068, 95% CI 2-sided [-0.308 to 0.443] — P-value, 95% CI, and estimated value are presented for Weeks 21-24

21. Secondary Outcome: Change From Baseline in Pain With Drinking Severity Scores
Description: Par. and/or parent/guardian recorded daily symptoms of eosinophilic esophagitis on a hand held personal digital assistant (electronic diary) during the Screening Phase, TP, and FP. A score of 6 was assigned the day participant did not drink. The severity of pain was assessed as: 1=didn't hurt at all, 2=hurt a little, 3=hurt somewhat, 4=hurt quite a bit, and 5=hurt a whole lot. The average difficulty and pain severity scores was calculated as the sum of the respective scores for that interval divided by the number of days in the interval. . Screening phase was considered as Baseline interval. Change from Baseline was calculated as the value for that interval minus the value for the Baseline interval. Analysis was performed using parametric ANCOVA models with terms for the relevant Baseline score, treatment group, age group and treatment by age group interaction.
Time Frame: Screening, Weeks 9-12 and Weeks 21-24
Population: as for outcome 13
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Scores on a scale
  Weeks 9-12, n=15,18,13 | -0.005 [-0.363 to 0.354] | 0.085 [-0.194 to 0.364] | -0.166 [-0.483 to 0.151]
  Weeks 21-24, n=13,16,11 | -0.193 [-0.734 to 0.347] | -0.006 [-0.384 to 0.372] | -0.118 [-0.591 to 0.356]
Statistical Analysis 1: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.691, ANCOVA; Mean Difference (Final Values) = 0.090, 95% CI 2-sided [-0.365 to 0.545] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 2: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.500, ANCOVA; Mean Difference (Final Values) = -0.161, 95% CI 2-sided [-0.639 to 0.317] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 3: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.568, ANCOVA; Mean Difference (Final Values) = 0.187, 95% CI 2-sided [-0.474 to 0.849] — P-value, 95% CI, and estimated value are presented for Weeks 21-24
Statistical Analysis 4: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.832, ANCOVA; Mean Difference (Final Values) = 0.076, 95% CI 2-sided [-0.643 to 0.794] — P-value, 95% CI, and estimated value are presented for Weeks 21-24

22. Secondary Outcome: Change From Baseline in Percentage of Days on Which the Participant Drank
Description: The percentage of days with the symptom of difficulty and pain when participant drank during each analysis interval (Baseline, Weeks 9-12 and Weeks 21-24) was calculated as the number of days the symptom was experienced divided by the number of days in the analysis interval, and presented as a percentage (ie, the proportion X 100%). Screening phase was considered as Baseline interval. Change from Baseline for each analysis interval was calculated as the value for that interval minus the value for the Baseline interval. Analysis was performed using parametric ANCOVA model with terms for Baseline score, treatment group, age group and treatment by age group interaction. The OC datasets with incorrect questionnaires excluded were used for the analysis.
Time Frame: Screening, Weeks 9-12 and Weeks 21-24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of days
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Percentage of days
  Weeks 9-12, n=15,18,13 | -0.24 [-2.27 to 1.80] | -1.08 [-2.61 to 0.45] | 0.66 [-1.06 to 2.39]
  Weeks 21-24, n=13,16,11 | -0.04 [-3.96 to 3.88] | -1.09 [-3.51 to 1.34] | -1.05 [-4.08 to 1.99]
Statistical Analysis 1: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.515, ANCOVA; Mean Difference (Final Values) = -0.85, 95% CI 2-sided [-3.45 to 1.76] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 2: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.496, ANCOVA; Mean Difference (Final Values) = 0.90, 95% CI 2-sided [-1.74 to 3.54] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 3: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.657, ANCOVA; Mean Difference (Final Values) = -1.05, 95% CI 2-sided [-5.82 to 3.72] — P-value, 95% CI, and estimated value are presented for Weeks 21-24
Statistical Analysis 4: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.691, ANCOVA; Mean Difference (Final Values) = -1.01, 95% CI 2-sided [-6.11 to 4.09] — P-value, 95% CI, and estimated value are presented for Weeks 21-24

23. Secondary Outcome: Change From Baseline in Difficulty With Eating Solid Foods
Description: Par. and/or parent/guardian recorded daily symptoms of eosinophilic esophagitis on a hand held personal digital assistant (electronic diary) during the Screening Phase, TP and FP. A score of 6 was assigned for that symptom when Par. did not eat solid foods. When Par.eat solid foods, the amount of difficulty was assessed as 1=no difficulty, 2=a little difficulty, 3=some difficulty, 4=quite a bit of difficulty, 5=a whole lot of difficulty. The average pain severity for the interval (Baseline, Weeks 9-12, Weeks 21-24) was calculated as the sum of the pain severity scores for that interval (including days assigned as 6) divided by the number of days in the interval. Screening phase was considered as Baseline interval. Change from Baseline was calculated as the value for that interval minus the value for the Baseline interval. Analysis was performed using parametric ANCOVA models with terms for the relevant Baseline score, treatment group, age group and treatment by age group interactions.
Time Frame: Screening, Weeks 9-12 and Weeks 21-24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Scores on a scale
  Weeks 9-12, n=15,18,13 | -0.474 [-0.794 to -0.153] | -0.174 [-0.422 to 0.074] | -0.119 [-0.418 to 0.180]
  Weeks 21-24, n=13,16,11 | -0.427 [-0.833 to -0.020] | -0.245 [-0.531 to 0.041] | -0.305 [-0.669 to 0.058]
Statistical Analysis 1: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.142, ANCOVA; Mean Difference (Final Values) = 0.300, 95% CI 2-sided [-0.105 to 0.704] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 2: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.115, ANCOVA; Mean Difference (Final Values) = 0.354, 95% CI 2-sided [-0.090 to 0.798] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 3: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.465, ANCOVA; Mean Difference (Final Values) = 0.182, 95% CI 2-sided [-0.319 to 0.683] — P-value, 95% CI, and estimated value are presented for Weeks 21-24
Statistical Analysis 4: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.649, ANCOVA; Mean Difference (Final Values) = 0.121, 95% CI 2-sided [-0.417 to 0.660] — P-value, 95% CI, and estimated value are presented for Weeks 21-24

24. Secondary Outcome: Change in Baseline in Pain With Eating Solid Foods Severity Scores
Description: Par. and/or parent/guardian recorded daily symptoms of eosinophilic esophagitis on a hand held personal digital assistant (electronic diary) during the Screening Phase, TP, and FP. A score of 6 was assigned for that symptom when Par. did not eat. The severity of pain was assessed when Par. eats food as: 1=didn't hurt at all, 2=hurt a little, 3=hurt somewhat, 4=hurt quite a bit, and 5=hurt a whole lot. The average pain severity for the interval (Baseline, Weeks 9-12, Weeks 21-24) was calculated as the sum of the pain severity scores for that interval (including days assigned as 6) divided by the number of days in the interval. Screening phase was considered as Baseline interval. Change from Baseline was calculated as the value for that interval minus the value for the Baseline interval. Analysis was performed using parametric ANCOVA models with terms for the relevant Baseline score, treatment group, age group and treatment by age group interaction.
Time Frame: Screening, Weeks 9-12 and Weeks 21-24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Scores on a scale
  Weeks 9-12, n=15,18,13 | -0.493 [-0.819 to -0.167] | -0.123 [-0.375 to 0.130] | -0.137 [-0.444 to 0.170]
  Weeks 21-24, n=13,16,11 | -0.399 [-0.900 to 0.102] | -0.109 [-0.462 to 0.244] | -0.271 [-0.724 to 0.182]
Statistical Analysis 1: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.077, ANCOVA; Mean Difference (Final Values) = 0.370, 95% CI 2-sided [-0.042 to 0.782] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 2: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.120, ANCOVA; Mean Difference (Final Values) = 0.356, 95% CI 2-sided [-0.097 to 0.809] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 3: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.345, ANCOVA; Mean Difference (Final Values) = 0.290, 95% CI 2-sided [-0.326 to 0.906] — P-value, 95% CI, and estimated value are presented for Weeks 21-24
Statistical Analysis 4: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.700, ANCOVA; Mean Difference (Final Values) = 0.128, 95% CI 2-sided [-0.541 to 0.798] — P-value, 95% CI, and estimated value are presented for Weeks 21-24

25. Secondary Outcome: Change From Baseline in the Percentage of Days Participants Ate Solid Foods
Description: The percentage of days with the symptom of difficulty and pain when eating solid foods during each analysis interval (Baseline, Weeks 9-12 and Weeks 21-24) was calculated as the number of days the symptom was experienced divided by the number of days in the analysis interval, and presented as a percentage (ie, the proportion X 100%). Screening phase was considered as Baseline interval. Change from Baseline for each analysis interval was calculated as the value for that interval minus the value for the Baseline interval. Analysis was performed using parametric ANCOVA model with terms for Baseline score, treatment group, age group and treatment by age group interaction. The OC datasets with incorrect questionnaires excluded were used for the analysis.
Time Frame: Screening, Weeks 9-12 and Weeks 21-24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of days
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Percentage of days
  Weeks 9-12, n=15,18,13 | 3.64 [-1.92 to 9.19] | 1.85 [-2.41 to 6.10] | 3.05 [-2.33 to 8.43]
  Weeks 21-24, n=13,16,11 | 2.26 [-2.69 to 7.21] | 0.65 [-2.84 to 4.14] | 1.81 [-3.11 to 6.72]
Statistical Analysis 1: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.609, ANCOVA; Mean Difference (Final Values) = -1.79, 95% CI 2-sided [-8.79 to 5.22] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 2: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.882, ANCOVA; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-8.55 to 7.38] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 3: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.595, ANCOVA; Mean Difference (Final Values) = -1.60, 95% CI 2-sided [-7.68 to 4.47] — P-value, 95% CI, and estimated value are presented for Weeks 21-24
Statistical Analysis 4: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.895, ANCOVA; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-7.34 to 6.44] — P-value, 95% CI, and estimated value are presented for Weeks 21-24

26. Secondary Outcome: Change From Baseline in Feeling of Something Stuck in Throat Bothersome Scores (for Par. 8-17 Years Only)
Description: Par. and/or parent/guardian recorded daily symptoms of the feeling like something is stuck in throat on a hand held personal digital assistant (electronic diary) during the Screening Phase, TP, and FP. A score of 0 was assigned for days on which the symptom of feeling of something stuck was not experienced. On days that feeling of something stuck in the throat was experienced, the amount the symptom bothered the Par. was assessed as 1=not bothered at all, 2=bothered a little, 3=somewhat bothered, 4=bothered quite a bit, 5=bothered a whole lot. Average bothersome score was calculated as the sum of the respective scores for that interval divided by the number of days. Screening phase was considered as Baseline interval. Change from Baseline was calculated as the value for that interval minus the value for the Baseline interval. Analysis was performed using parametric ANCOVA models with terms for the relevant Baseline score, treatment group, age group and treatment by age interaction.
Time Frame: Screening, Weeks 9-12 and Weeks 21-24
Population: as for outcome 16
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Scores on a Scale
  Weeks 9-12, n=12,12,8 | -0.751 [-1.135 to -0.368] | -0.238 [-0.621 to 0.145] | -0.510 [-0.982 to -0.038]
  Weeks 21-24, n=11,11,8 | -0.785 [-1.354 to -0.216] | -0.075 [-0.646 to 0.496] | -0.535 [-1.207 to 0.137]
Statistical Analysis 1: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.062, ANCOVA; Mean Difference (Final Values) = 0.513, 95% CI 2-sided [-0.028 to 1.055] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 2: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.425, ANCOVA; Mean Difference (Final Values) = 0.241, 95% CI 2-sided [-0.369 to 0.852] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 3: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.082, ANCOVA; Mean Difference (Final Values) = 0.710, 95% CI 2-sided [-0.096 to 1.516] — P-value, 95% CI, and estimated value are presented for Weeks 21-24
Statistical Analysis 4: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.564, ANCOVA; Mean Difference (Final Values) = 0.250, 95% CI 2-sided [-0.631 to 1.132] — P-value, 95% CI, and estimated value are presented for Weeks 21-24

27. Secondary Outcome: Change From Baseline in Percentage of Days With Feeling of Something Stuck in Throat (for Par. 8-17 Years)
Description: The percentage of days with feeling of something stuck in throat during each analysis period (Baseline, Weeks 9-12 and Weeks 21-24) was calculated as the number of days the symptom was experienced divided by the number of days in the analysis interval, and presented as a percentage (ie, the proportion X 100%). Screening phase was considered as Baseline interval. Change from Baseline for each analysis interval was calculated as the value for that interval minus the value for the Baseline interval. Analysis was performed using parametric ANCOVA model with terms for Baseline score, treatment group, age group and treatment by age group interaction. The OC datasets with incorrect questionnaires excluded were used for the analysis.
Time Frame: Screening, Weeks 9-12 and Weeks 21-24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of days
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Percentage of days
  Weeks 9-12, n=12,12,8 | -21.56 [-33.73 to -9.40] | -12.11 [-24.29 to 0.06] | -17.44 [-32.34 to -2.54]
  Weeks 21-24, n=11,11,8 | -21.33 [-38.48 to -4.17] | -10.76 [-27.95 to 6.42] | -15.84 [-35.89 to 4.22]
Statistical Analysis 1: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.270, ANCOVA; Mean Difference (Final Values) = 9.45, 95% CI 2-sided [-7.77 to 26.67] — P-value, 95% CI, and estimated value are presented for Weeks 9-12
Statistical Analysis 2: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.664, ANCOVA; Mean Difference (Final Values) = 4.12, 95% CI 2-sided [-15.11 to 23.36] — P-value, 95% CI, and estimated value are presented for Weeks 21-24
Statistical Analysis 3: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.381, ANCOVA; Mean Difference (Final Values) = 10.57, 95% CI 2-sided [-13.81 to 34.94] — P-value, 95% CI, and estimated value are presented for Weeks 21-24
Statistical Analysis 4: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.672, ANCOVA; Mean Difference (Final Values) = 5.49, 95% CI 2-sided [-20.87 to 31.86] — P-value, 95% CI, and estimated value are presented for Weeks 21-24

28. Secondary Outcome: Number of Participants With Maintenance of Response
Description: Participants who achieved a response of <5 esophageal eosinophils/HPF at Week 12 by worst case analysis, were evaluated for maintenance of response of <20 cells/HPF at Week 24. Response categories were defined as: non-responder (did not respond at Week 12 or Week 24); delayed responder (did not respond at Week 12 but responded at Week 24); relapsed (responded at Week 12 but not at Week 24); maintained (responded at Week 12 and Week 24). The following assumptions were made for worst case: if a Participant dropped out of the study due to lack of efficacy or an adverse event and had a missing response, their response was imputed as not achieved (i.e. failure). However for Participants withdrawn for other reasons (e.g. lost to follow-up) with a missing response (i.e. did not have the biopsy) the response was made as missing and not imputed.
Time Frame: Week 12 and Week 24
Population: ITT Population. Only those participants were responders at Week 12 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 16 | 20 | 20
Participants
  Non-responder | 12 | 18 | 18
  Delayed responder | 1 | 0 | 2
  Relapsed | 2 | 1 | 0
  Maintained | 1 | 1 | 0
Statistical Analysis 1: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.400, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.111, Cochran-Mantel-Haenszel

29. Secondary Outcome: Mean Change From Baseline in Peak Esophageal Eosinophil Counts at Weeks 12 and 24
Description: Participants underwent an esophagogastroduodenoscopy (EGD) with biopsies at Screening and at Weeks 12 and 24. Peak esophageal eosinophils were calculated as the maximum count across all esophageal biopsies at each time point. Screening value was considered as the Baseline value. Change from baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Cells/HPF
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Cells/HPF
  Week 12, n=17,20,20 | -76.8 (16.13) | -95.2 (19.63) | -78.9 (13.62)
  Week 24, n=16,19,19 | -26.3 (16.52) | -41.6 (23.71) | -60.1 (15.01)
Statistical Analysis 1: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.421, van Elteren test; Mean Difference (Final Values) = -18.3, 95% CI 2-sided [-71.1 to 34.4] — P-value, 95% CI, and Estimated value are presented for Change from Baseline at Week 12
Statistical Analysis 2: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.633, van Elteren test; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-44.6 to 40.5] — P-value, 95% CI, and Estimated value are presented for Change from Baseline at Week 12
Statistical Analysis 3: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.920, van Elteren test; Mean Difference (Final Values) = -15.3, 95% CI 2-sided [-76.3 to 45.7] — P-value, 95% CI, and Estimated value are presented for Change from Baseline at Week 24
Statistical Analysis 4: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.105, van Elteren test; Mean Difference (Final Values) = -33.8, 95% CI 2-sided [-79.2 to 11.6] — P-value, 95% CI, and Estimated value are presented for Change from Baseline at Week 24

30. Secondary Outcome: Change From Baseline in Mean Esophageal Eosinophil Counts at Weeks 12 and 24
Description: Participants underwent an EGD with biopsies at Screening and at Weeks 12 and 24. Mean esophageal eosinophils were calculated as the mean number across all esophageal biopsies at each time point. Screening value was considered as the Baseline value. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Cells/HPF
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Cells/HPF
  Week 12, n=17,20,20 | -27.34 (6.323) | -29.97 (6.184) | -34.04 (5.984)
  Week 24, n=16, 19, 19 | -8.23 (6.449) | -17.48 (7.446) | -26.03 (5.677)
Statistical Analysis 1: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.747, van Elteren test; Mean Difference (Final Values) = -2.63, 95% CI 2-sided [-20.68 to 15.41] — P-value, 95% CI, and Estimated value are presented for change from baseline values at Week 12
Statistical Analysis 2: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.352, van Elteren test; Mean Difference (Final Values) = -6.70, 95% CI 2-sided [-24.41 to 11.01] — P-value, 95% CI, and Estimated value are presented for change from baseline values at Week 12
Statistical Analysis 3: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 2.5 mg/kg; Test type: Superiority or Other; p = 0.525, van Elteren test; Mean Difference (Final Values) = -9.25, 95% CI 2-sided [-29.69 to 11.20] — P-value, 95% CI, and Estimated value are presented for change from baseline values at Week 24
Statistical Analysis 4: Comparison: Mepolizumab 0.55 mg/kg vs Mepolizumab 10 mg/kg; Test type: Superiority or Other; p = 0.071, Van Elteren test; Mean Difference (Final Values) = -17.79, 95% CI 2-sided [-35.21 to -0.38] — P-value, 95% CI, and Estimated value are presented for change from baseline at week 24

31. Secondary Outcome: Absolute Blood Eosinophils Count at the Indicated Time Points
Description: Blood samples were obtained at Screening, pre-infusion and 24h and 72-96h post-infusion at Day 1, Weeks 4 and 8; and at Week 2, 6, 10, 12, 16, 20, 24 and 34 visits or Early Withdrawal Visit to estimate blood eosinophil count.
Time Frame: Screening, Day 1, Weeks 2, 4, 6, 8, 10, 12, 16, 20, 24 and 34
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Giga cells per liter (GI/L)
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Giga cells per liter (GI/L)
  Screening, n=17,16,20 | 0.441 (0.2358) | 0.524 (0.2579) | 0.493 (0.2218)
  Day 1 predose, n= 17,19,20 | 0.419 (0.1620) | 0.476 (0.2660) | 0.559 (0.2987)
  Day 1 24h postdose, n=12,10,14 | 0.147 (0.0623) | 0.158 (0.1156) | 0.230 (0.1120)
  Day 1 72-96h postdose, n=14,11,11 | 0.123 (0.0930) | 0.151 (0.0823) | 0.179 (0.1319)
  Week 2, n=19,18,20 | 0.139 (0.1531) | 0.114 (0.0815) | 0.111 (0.068)
  Week 4 predose, n=19,16,20 | 0.165 (0.1635) | 0.072 (0.0571) | 0.062 (0.0381)
  Week 4 24h postdose, n=16,14,14 | 0.093 (0.0690) | 0.097 (0.0548) | 0.079 (0.0285)
  Week 4 72-96h postdose, n=15,15,15 | 0.081 (0.0666) | 0.089 (0.0721) | 0.053 (0.0377)
  Week 6, n=19,16,20 | 0.099 (0.0897) | 0.060 (0.0678) | 0.146 (0.3902)
  Week 8 predose, n=19,19,19 | 0.113 (0.0910) | 0.081 (0.0517) | 0.052 (0.0385)
  Week 8 24h postdose, n=17,14,14 | 0.077 (0.0645) | 0.055 (0.0494) | 0.061 (0.0305)
  Week 8 72-96h postdose, n= 16,15,13 | 0.070 (0.0803) | 0.045 (0.0566) | 0.075 (0.0285)
  Week 10, n= 18,18,18 | 0.100 (0.0872) | 0.059 (0.0537) | 0.043 (0.0412)
  Week 12, n=16,18,20 | 0.091 (0.0686) | 0.070 (0.1116) | 0.048 (0.0411)
  Week 16, n=15,18,19 | 0.261 (0.2097) | 0.076 (0.0619) | 0.078 (0.0517)
  Week 20, n=15,17,18 | 0.478 (0.3944) | 0.191 (0.0893) | 0.124 (0.0658)
  Week 24, n=15,20,18 | 0.706 (0.4513) | 0.389 (0.2756) | 0.147 (0.1167)
  Week 34, n=14,18,16 | 0.650 (0.3025) | 0.569 (0.2599) | 0.575 (0.4268)

32. Secondary Outcome: Plasma Concentration of Mepolizumab
Description: Blood samples were obtained at pre-infusion and 5m, 2h, 24h, 72-96h post-infusion at Day 1, Weeks 4, 8; and Weeks 2, 6 10, 12, 16, 20, 24 and 34 to estimate the plasma concentration of mepolizumab. Only those participants available at specified time points are analyzed (represented as n=X,X,X in the category titles).
Time Frame: Day 1, Weeks 2, 4, 6, 8, 10, 12, 16, 20, 24 and 34
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Microgram per milliliter (µg/mL)
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Number analyzed (Participants) | 19 | 20 | 20
Microgram per milliliter (µg/mL)
  Day 1 5mins postdose, n=18,20,19 | 11.3 (7.172) | 39.56 (19.041) | 177.94 (70.581)
  Day 1 2h postdose, n=18,19,17 | 11.34 (3.516) | 42.38 (14.895) | 192.99 (49.243)
  Day 1 24h postdose, n=18,19,16 | 8.32 (2.428) | 30.05 (7.974) | 144.26 (43.87)
  Day 1 72-96h postdose, n=15,19,17 | 6.08 (1.907) | 22.62 (7.306) | 111.87 (30.046)
  Week 2, n=17,16,18 | 3.42 (1.381) | 16.08 (4.68) | 59.2 (16.636)
  Week 4 Predose,n=19,20,19 | 1.83 (0.643) | 9.43 (2.884) | 37.29 (21.978)
  Week 4, 5 min postdose, n=19,19,18 | 9.69 (3.097) | 61.56 (18.021) | 204.93 (69.325)
  Week 4 2h postdose, n=19,19,20 | 10.04 (3.241) | 50.75 (12.992) | 212.5 (71.48)
  Week 4 24h postdose, n=19,15,20 | 8.07 (2.515) | 42.89 (11.337) | 189.92 (55.81)
  Week 4, 72-96h postdose, n=19,18,17 | 6.35 (2.497) | 34.54 (8.188) | 143.47 (38.414)
  Week 6, n=17,13,17 | 3.69 (1.031) | 20.13 (6.602) | 88.14 (42.311)
  Week 8 predose, n=17,16,16 | 2.48 (0.69) | 10.97 (4.072) | 50.96 (17.244)
  Week 8 5 min postdose, n=19,20,18 | 12.44 (3.285) | 57.3 (18.132) | 213.05 (51.882)
  Week 8 2h postdose, n=19,19,19 | 12.45 (3.386) | 58.28 (16.981) | 217.71 (51.983)
  Week 8 24 h postdose, n=18,18,17 | 9 (2.554) | 47.13 (12.09) | 173.41 (43.848)
  Week 8 72-96h postdose, n=17,19,19 | 6.89 (1.651) | 36.49 (11.133) | 145.75 (35.48)
  Week 10, n=19,15,16 | 4.56 (1.192) | 20.7 (6.977) | 90.38 (26.77)
  Week 12, n=14,18,15 | 2.57 (0.965) | 11.19 (3.395) | 48.8 (20.314)
  Week 16, n=14,16,17 | 0.79 (0.474) | 4.04 (1.768) | 16.38 (6.523)
  Week 20, n=11,14,15 | 0.27 (0.16) | 1.27 (0.535) | 5.76 (2.477)
  Week 24, n=8,14,12 | 0.11 (0.056) | 0.67 (0.389) | 2.13 (2.368)
  Week 34, n=1,5,7 | 0.06 (NA) — There were too few participants to provide a dispersion value. | 0.08 (0.025) | 1.14 (1.882)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the date of the first dose of study medication up to the Week 12.
Description: AEs and SAEs were collected in the members of ITT Population, comprised of all participants in the treatment cohort who gave informed consent, were randomized and received at least one dose of study medication.
Arm/Group | Mepolizumab 0.55 mg/kg | Mepolizumab 2.5 mg/kg | Mepolizumab 10 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/19 | 1/20 | 2/20
Other Adverse Events (participants affected / at risk) | 18/19 | 14/20 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mepolizumab 0.55 mg/kg (N=19) | Mepolizumab 2.5 mg/kg (N=20) | Mepolizumab 10 mg/kg (N=20)
Foreign body trauma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Oesophageal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mepolizumab 0.55 mg/kg (N=19) | Mepolizumab 2.5 mg/kg (N=20) | Mepolizumab 10 mg/kg (N=20)
Any event (Gastrointestinal disorders) | 10 | 8 | 7
Vomiting (Gastrointestinal disorders) | 5 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 3
Nausea (Gastrointestinal disorders) | 4 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Eosinophilic oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Any event (Infections and infestations) | 10 | 7 | 8
Nasopharyngitis (Infections and infestations) | 5 | 1 | 4
Ear infection (Infections and infestations) | 1 | 1 | 1
Influenza (Infections and infestations) | 1 | 2 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 1 | 1
Sinusitis (Infections and infestations) | 2 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 2
Otitis media (Infections and infestations) | 2 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Eczema infected (Infections and infestations) | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0
Orchitis (Infections and infestations) | 1 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Any event (Respiratory, thoracic and mediastinal disorders) | 9 | 7 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Any event (Nervous system disorders) | 6 | 2 | 6
Headache (Nervous system disorders) | 2 | 2 | 4
Dizziness (Nervous system disorders) | 1 | 0 | 2
Aphonia (Nervous system disorders) | 1 | 0 | 0
Hypersomnia (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0 | 0
Any event (General disorders) | 5 | 0 | 5
Pyrexia (General disorders) | 4 | 0 | 2
Chest pain (General disorders) | 0 | 0 | 2
Catheter site pain (General disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0
Granuloma (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 0
Peripheral coldness (General disorders) | 0 | 0 | 1
Any event (Skin and subcutaneous tissue disorders) | 6 | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Any event (Injury, poisoning and procedural complications) | 3 | 3 | 2
Joint sprain (Injury, poisoning and procedural complications) | 1 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foreign body trauma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Oesophageal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 1
Any event (Immune system disorders) | 0 | 2 | 3
Seasonal allergy (Immune system disorders) | 0 | 0 | 2
Food allergy (Immune system disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Multiple allergies (Immune system disorders) | 0 | 1 | 0
Any event (Renal and urinary disorders) | 1 | 1 | 2
Dysuria (Renal and urinary disorders) | 1 | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Any event (Eye disorders) | 1 | 0 | 2
Conjunctivitis (Eye disorders) | 0 | 0 | 1
Eye irritation (Eye disorders) | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1
Any event (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Any event (Blood and lymphatic system disorders) | 2 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0 | 0
Any event (Psychiatric disorders) | 0 | 1 | 1
Aggression (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Any event (Reproductive system and breast disorders) | 2 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 1 | 0 | 0
Any event (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Any event (Hepatobiliary disorders) | 0 | 1 | 0
Hyperbilirubinuria (Hepatobiliary disorders) | 0 | 1 | 0
Any event (Investigations) | 1 | 0 | 0
Blood urine present (Investigations) | 1 | 0 | 0
Any event (Metabolism and nutrition disorders) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Any event (Vascular disorders) | 1 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.